CLINICAL TRIAL: NCT03146611
Title: Neutrophil CD64 Versus Neutrophil/Lymphocyte Ratio (NLR) as Markers Predicting In-hospital Outcome in Acute Exacerbation of COPD
Brief Title: nCD64 vs. Neutrophil/Lymphocyte Ratio for Predicting In-hospital Outcome in AE-COPD
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Prof. Dr. Aliae AR Mohamed-Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU5
Record Dates: First submitted 2017-04-22; First posted 2017-05-10 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: COPD Exacerbation; Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients: A diagnosis of COPD was made by a clinical history, examination and spirometer (forced expiratory volume in 1st second/forced vital capacity (FEV1/FVC)ratio of <0.7). The severity of COPD was graded according to the Global Initiative for Chronic Obstructive Lung Disease guidelines. [9] (Stage I, mild COPD: FEV1≥80.0% predicted; Stage II, moderate COPD: FEV1 80-50.0%; Stage III, severe COPD: FEV1 50- 30.0%; Stage IV, very severe COPD: FEV1< 30.0%). The exacerbation of COPD was defined as the patient being diagnosed with COPD with two or more of the following three symptoms of exacerbations: new or worsening cough, worsened dyspnea, and worsened sputum volume and/or change in its color.
  Interventions: Diagnostic Test: nCD64; Diagnostic Test: Neutrophil/Lymphocyte Ratio
- control: healthy sex and age matched group
  Interventions: Diagnostic Test: nCD64; Diagnostic Test: Neutrophil/Lymphocyte Ratio

INTERVENTIONS:
Diagnostic Test: nCD64 — neutrophil CD64
  Other Names: neutrophil CD64
Diagnostic Test: Neutrophil/Lymphocyte Ratio — Neutrophil/ lymphocyte ratio
  Other Names: NLR

SUMMARY:
Neutrophil CD64 versus Neutrophil/Lymphocyte ratio (NLR) as markers predicting in-hospital outcome in acute exacerbation of COPD

DETAILED DESCRIPTION:
Acute exacerbation of COPD is among the most frequent reasons for hospitalisation. Approximately 4% of the general population in the western world is admitted with an acute respiratory disease at least once a year and nearly one fifth of hospital visits is due to acute exacerbation of COPD. Early identiﬁcations and management of AE-COPD is an important issue in clinical practice. AE-COPD is accompanied with various worsening respiratory symptoms and deterioration in lung function. Also the frequency and severity of attacks is associated with increased mortality.

During exacerbation, the inﬂammation in COPD is ampliﬁed in comparison with stable periods. The increased level of inﬂammatory markers is associated with lung function decline. As infection, is the main cause leading to clinical AECOPD, white blood cell counts and ESR are the common markers to show the existence of infection in patients with COPD. Recently, other bio markers are used. Authors have found that the high-affinity Fc receptor-CD64 is expressed by monocytes and only weakly on resting neutrophils. The high-expression of neutrophil CD64 (nCD64) is an early step in the host- immune response to bacterial infection. Studies have shown that the nCD64 might be used as a bio-marker for early-onset sepsis or bacterial infection. However, authors agreed that the value of the nCD64 in COPD prognosis is unknown.

As most of novel bio-markers that identify the severity of acute exacerbation in COPD, are time consuming and expensive, there is a need to use more simple tests. The Neutrophil-lymphocyte ratio is a rapid, easy and cost-effective method derived from routine complete blood count tests in clinical practice. The NLR could be an important marker that assess inﬂammatory status in patients with COPD and could identify early, acute exacerbation. However, this bio marker has not been widely used in the diagnosis of AECOPD.

The purpose of the present study is: 1- To measure the values of the neutrophil CD64 and NLR in patients with AECOPD and stable COPD, 2- to correlate between nCD64, NLR and the usual routine bio-markers as white blood cell count and erythrocyte sedimentation rate, 3- to investigate the role of nCD64 and NLR as predictors for short term hospital outcome in this group.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as AECOPD and stable COPD ( random selection by 1:1 cross over). A diagnosis of COPD was made by a clinical history, examination and spirometer (forced expiratory volume in 1st second/forced vital capacity (FEV1/FVC)ratio of <0.7). The severity of COPD was graded according to the Global Initiative for Chronic Obstructive Lung Disease guidelines.

Exclusion Criteria:

* history of current respiratory disorders other than COPD, malignancy, systemic auto-immune disorders, recent surgery and severe endocrine, hepatic or renal diseases. Patients with pneumonia, cardiovascular and metabolic diseases

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The exacerbation of COPD is defined as the patient being diagnosed with COPD with two or more of the following three symptoms of exacerbations: new or worsening cough, worsened dyspnea, and worsened sputum volume and/or change in its color.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Define the cut off values of the nCD64 and NLR in patients with AE-COPD and stable COPD | 3 months
  level of nCD64 and NLR that define exacerbation

SECONDARY OUTCOMES:
Can nCD64 and NLR as markers be used as predictors for short term hospital outcome | 3 months
  correlate between level of these markers and hospital outcome

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No